CLINICAL TRIAL: NCT05473871
Title: Enhancing Capacity in Faith-based Organizations to Implement and Sustain Multilevel Innovations to Improve Physical Activity
Brief Title: Enhancing Capacity in Churches to Implement PA Programs
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: San Diego State University (Other)
Collaborators: Washington University School of Medicine (Other); University of California, Berkeley (Other); University of California, San Diego (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: HS-2020-0221; R01HL158538 (NIH)
Record Dates: First submitted 2022-07-21; First posted 2022-07-26 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Cardiovascular Diseases
Keywords: Physical Activity; Faith in Action; Hispanic Women; Latinas; Exercise
MeSH Terms: conditions — Cardiovascular Diseases; Motor Activity

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Triple
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard EBI Condition (Experimental): Faith in Action as originally implemented
  Interventions: Behavioral: Faith in Action
- Enhanced Condition (Experimental): Standard condition + organizational-level implementation strategies
  Interventions: Behavioral: Faith in Action+
- Enhanced + Sustainment condition (Experimental): Enhanced implementation condition + maintenance strategies
  Interventions: Behavioral: Faith in Action++

INTERVENTIONS:
Behavioral: Faith in Action — Interpersonal level: Group exercise classes offered 6 days/week (walking, cardio dance, strength training), Kickoff event
  Individual level: Motivational Interviewing calls every 6 months, Health handouts on 14 topics distributed at PA classes
  Arms: Standard EBI Condition
Behavioral: Faith in Action+ — Standard Faith in Action Intervention plus: 1) Health Behavior Change Workshop for FBO leaders; 2) Targeted Messaging; and 3) Empowerment Training for Promotoras
  Arms: Enhanced Condition
Behavioral: Faith in Action++ — Enhanced Condition plus: 1) Foster community collaborations and 2) Provide maintenance support
  Arms: Enhanced + Sustainment condition

SUMMARY:
Despite the benefits of physical activity (PA) to prevent cardiovascular disease and other chronic diseases, few adult Latinas meet PA guidelines. Given the central role of churches within the Latino community and their commitment to the well-being of their members, they are ideal settings for health promotion. Evidence-based interventions (EBIs) for increasing PA and reducing obesity exist, but few PA interventions go to scale. Investigators propose to enhance Faith in Action with three organization-level strategies designed to increase program fit and effectiveness: 1) training church leaders in health promotion; 2) tailoring messaging to enhance fit between Faith in Action and each unique church environment; and 3) empowering community health workers (promotoras) to advocate for organizational change. Given the need to improve strategies to sustain health programs in community settings, investigators will test the influence of two additional sustainment strategies: 1) strengthening community collaborations and 2) providing technical support. Thirty-two churches will be randomly assigned to a Standard EBI group (Faith in Action as originally implemented), an Enhanced group (Standard intervention + organizational-level implementation strategies), or an Enhanced + Sustainment group (Enhanced implementation group + sustainment strategies). Investigators will test the proposed implementation strategies on organization-level change and individual behavior in diverse churches for a 12-month intervention and 6-month follow-up period. The proposed study aims to: 1) Test the short and long-term impacts of organization-level implementation strategies in 2 Enhanced conditions on organizational outcomes compared to the Standard EBI condition and 2) Examine individual behavior change among Latinas (N=677) in churches in the 2 Enhanced conditions compared to the Standard EBI condition. The study's primary hypothesis is that Latina's receiving the Enhanced interventions will increase their PA levels significantly more than those receiving the Standard Faith in Action intervention, and the improvements in PA will be sustained. If successful, findings from the current study will provide evidence of organizational-level strategies for uptake, sustainment, and implementation strategies for scale-up of PA interventions to increase PA and reduce chronic disease in churches across the US.

DETAILED DESCRIPTION:
This study, guided by PRISM/RE-AIM frameworks, will use a pragmatic, cluster randomized controlled design to stratify by faith-based organization (FBO) size, and randomly assign 32 FBOs to one of 3 conditions: a Standard implementation condition (n=8 FBOs), an Enhanced implementation condition (Standard + organizational implementation strategies; n=12 FBOs), or an Enhanced + Sustainment condition (Enhanced + sustainment strategies; n=12 FBOs) for a 12-mo intervention with a 6-month sustainment follow- up period. This design offers the opportunity to examine the impact of explicit implementation and sustainment strategies compared to the Standard EBI condition to advance the science on scaling up EBIs. Investigators will allocate more churches in the Enhanced conditions to provide more opportunities to test the implementation process and impact of the proposed strategies in diverse church contexts. This design will allow investigators to examine the additive impact of the organization-level implementation strategies on both organizational outcomes (Aim 1) and individual outcomes (Aim 2). Investigators will examine the potential mechanisms of action (Secondary Aim 1) of the organizational implementation strategies. At 12 months post-baseline, FBOs in the Standard (n=8) and Enhanced condition (n=12) will receive no additional support while FBOs in the Enhanced + Sustainment condition (n=12) will receive additional program support (Secondary Aim 2) to examine the impact of sustainment strategies on both program and participant PA sustainment over an additional 6 months. Quantitative and qualitative data will be collected at baseline, 6 months, 12 months, and 18 months post baseline.

ELIGIBILITY:
Inclusion Criteria:

* Self-identifying as Latina
* Aged 18-65 years
* Planning on attending the FBO for the next 18 months
* Low self-reported leisure-time MVPA (<50 min of weekly leisure MVPA)
* No health factors interfering with PA

Exclusion Criteria:

* Anyone with a health condition precluding them from engaging in PA
* Cognitive impairment preventing participation
* Inability to complete the informed consent in English or Spanish
* Attending other churches besides the church of recruitment

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 677 (Estimated)
Dates: Start 2022-11-15 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Organizational Level: Change in Innovation-Values fit from Baseline to Month 6 | 6 months
  Investigators will survey FBO leaders, church staff, promotoras, and parishioners to assess the change in Innovation-values fit from baseline to month 6. Self-report questions regarding perceptions of the fit between the values of their FBO and the Faith in Action intervention will be measured using Likert scales (completely agree to completely disagree).
Organizational Level: Change in Innovation-Values fit from Baseline to Month 12 | 12 months
  Investigators will survey FBO leaders, church staff, promotoras, and parishioners to assess the change in Innovation-values fit from baseline to month 12. Self-report questions regarding perceptions of the fit between the values of their FBO and the Faith in Action intervention will be measured using Likert scales (completely agree to completely disagree).
Individual Level: Change in Participants' Moderate to Vigorous Physical Activity (MVPA) from Baseline to Month 6 | 6 months
  Investigators will assess the change in the number of minutes per day of participants' MVPA from baseline to month 6.
Individual Level: Change in Participants' Moderate to Vigorous Physical Activity (MVPA) from Baseline to Month 12 | 12 months
  Investigators will assess the change in the number of minutes per day of participants' MVPA from baseline to month 12.

SECONDARY OUTCOMES:
Organizational Level: Maintenance of Promotoras' PA Class Delivery | 18 months post-baseline
  Investigators will assess if the promotoras are delivering at least 3 PA classes per week at their church.
Organizational Level: Maintenance of Promotoras' MI Calls | 18 months post-baseline
  Investigators will assess if promotoras have made at least 1 MI call.
Individual Level: Maintenance of Moderate to Vigorous Physical Activity (MVPA) at 18 months | 18 months post-baseline
  Investigators will compare the number of minutes of participants' MVPA per day at 18 months to baseline, 6, and 12 months, to assess maintenance of MVPA at 18 months, which will be 6 months after the intervention has ended.

CONTACTS AND LOCATIONS:
Overall Officials: Elva Arredondo, PhD, Principal Investigator — San Diego State University
Locations (1):
- San Diego State University Research Foundation, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: Yes
The final dataset will be an electronic database containing objective (BMI and Blood Pressure) and self-report (survey with primary and secondary outcomes, demographic information, etc.) variables from baseline, 6, 12, and 18 months. Data will be de-identified to remove all subject identifiers.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will become available after initial data analyses and preparation of major publications.
Access Criteria: Researchers interested in accessing the data must complete a registration process and must agree to the conditions of use, including restrictions against attempting to identify study participants, destruction of the data after analyses are completed, reporting responsibilities, restrictions on redistribution of the data to third parties, and proper acknowledgement of the data resource. Those interested in accessing data must submit a brief proposal describing the intended use of the data; the investigative team will determine the scientific soundness of the proposal, as well as whether adequate data protections in place, as part of the decision for the researcher to be able to access the dataset.